CLINICAL TRIAL: NCT00842283
Title: Role of Angiogenesis in Dermatologic Diseases: A Potential Therapeutic Target
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Kristen Kelly, Professor of Dermatology, University of California, Irvine
Other Study IDs: 20076094
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Dermatologic Diseases
Keywords: dermatologic diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- dermatologic diseases: skin tissue sample
  Interventions: Other: skin tissue sample

INTERVENTIONS:
Other: skin tissue sample — skin tissue sample

SUMMARY:
The researchers believe that pro-angiogenic factors are upregulated in a wide range of dermatologic diseases, including port wine stains, hemangiomas, angiofibromas, Kaposi's sarcoma, angiosarcoma, scars, rosacea, and psoriasis. Select specimens may undergo genetic analysis to investigate underlying molecular pathways associated with dysregulated angiogenesis in cutaneous disease.

Biospecimens, either previously obtained or newly collected from dermatologic conditions, will be analyzed for angiogenic markers. Discarded skin tissue from surgical or biopsy procedures may also be used, including both diseased and non-diseased tissue from the same donor. Some specimens may also undergo genetic analysis to investigate underlying molecular pathways.

De-identified data such as age, sex, race, cause of death, lesion location, and description will be recorded. Currently, specimens are limited to clinically diagnosed lesions not typically biopsied, or lesions already confirmed by prior biopsy.

DETAILED DESCRIPTION:
Biospecimens from various dermatologic diseases, including port wine stains, hemangiomas, angiofibromas, Kaposi's sarcoma, angiosarcoma, scars, rosacea, and psoriasis will be evaluated for markers of angiogenesis. Additionally, researchers can use discarded human skin tissue samples from skin biopsy/surgery sites, which are removed for closure but are not submitted for histopathologic analysis. We may use donated tissue with both dermatologic disease and non-diseased tissue from the same donor. Biopsies may also be taken for molecular and genetic analysis of specimen. Non-identifiable information regarding the patient, such as age, sex, race, cause of death, location, and description of diseased skin may be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older.
* willing to have a skin biopsy

Exclusion Criteria:

* under 16 years of age
* unable to carry out instructions

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Tissue samples will be collected from Dermatopathology Lab, Pathology lab, discarded tissue from dermatologic surgery at University of California Irvine. Additional biopsies may be obtained of known lesions.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2008-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Factors in dermatologic diseases. | up to 4 weeks
  Evaluate the role of angiogenesis in cutaneous disease and ultimately, facilitate implementation of anti-angiogenic therapy in a wide range of dermatologic diseases including port wine stains, hemangiomas, angiofibromas, Kaposi's sarcoma, angiosarcoma, scars, rosacea and psoriasis.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelly, MD, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - Beckman Laser Institute and Medical Clinic, Irvine, California
  - Dermatology Clinic at Gavin Herbert Eye Institute, Irvine, California

IPD SHARING:
Plan to Share IPD: No